CLINICAL TRIAL: NCT01629108
Title: Normative Values in Audiovestibular Testing
Brief Title: Normal Values in Hearing and Balance Testing
Status: Recruiting | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120152; 12-DC-0152
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-08-14

CONDITIONS: Healthy Volunteer
Keywords: Normative Data; Vestibular; Auditory; Healthy Volunteers; Hearing; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy volunteers aged 5 to 80

SUMMARY:
Background:

- Researchers at the National Institutes of Health give many tests of hearing and balance. These tests can help detect problems that affect hearing or balance. It is important to know exactly how healthy people perform on each of these tests. This information will indicate when a test result is normal and when a test result shows a problem. Researchers also want to determine the best methods for each test.

Objectives:

- To test different types of hearing and balance tests, and collect information on normal values for each test.

Eligibility:

- Healthy volunteers between 5 and 80 years of age.

Design:

* This study will require a single visit to the National Institutes of Health Clinical Center. It will include both screening tests and study tests of hearing and balance. Sometimes, a second visit may be required if a test is designed to measure the same thing on 2 different days. Each visit will last between 2 and 5 hours, depending on the number of tests scheduled per visit.
* Participants will have a physical exam and medical history. They will also have basic tests to check for normal hearing and balance.
* Participants may have different hearing tests, including the following:
* Auditory Evoked Potentials to study how the ears and brain handle sound information.
* Auditory Processing Tests to study how a person processes complex sounds like speech in background noise.
* Tests of middle ear and inner ear function.
* Participants may have different balance and inner ear tests, including the following:
* Balance test on a tilting platform.
* Different tests to measure how well the eyes, ears, and brain work together to help maintain balance.
* Treatment will not be needed as part of this study.

DETAILED DESCRIPTION:
Objective:

This is a normative data collection protocol. The primary objective is to establish the normative range of data for the NIH research population on tests of auditory and vestibular function that employ parameters and/or methodologies that are either new or unique to the NIH, have been upgraded (software and/or hardware), or have not been well standardized in the literature. Use of the normative data will be two-fold: 1) it will serve as a reference interval of normal performance by which test results can be interpreted as normal or abnormal and, in some cases 2) it will be used as control data for the purpose of comparison to data obtained in various patient groups.

Secondary objectives, when applicable, are to evaluate: 1) the effect of a change in methodology, stimulus characteristics, test equipment, or test paradigm on normative data for existing measures, 2) the influence of subject age and gender on normative data, and 3) intra-subject variability on repeated measures.

This protocol provides the construct for small, targeted normative studies and, subsequently, there are no specific a priori hypotheses.

Study population:

Healthy volunteers ranging in age from 5-80 years will be studied under this protocol.

Design:

This protocol is designed to collect normative data on tests of audiometric and vestibular function. Small study tasks will be conducted on healthy volunteers in order to determine the normal distribution of performance on defined subsets of hearing and/or balance tests. These study tasks will fall into one of the following five general categories: serial monitoring of auditory function, auditory evoked potentials, auditory processing, middle ear function, and vestibular function. All participants will have a basic hearing test and tympanometry to confirm eligibility for the protocol. The subsequent measures of auditory or vestibular function will depend on the defined subset of tests for which normative data is being sought. Possible tests for normal data collection would include: middle ear function tests (MEF), otoacoustic emissions (OAE), auditory evoked potentials (AEP), tests of auditory processing (AP), computerized dynamic platform posturography (CDPP), vestibular evoked myogenic potentials (VEMP), videonystagmography (VNG) and/or rotational vestibular testing (RVT).

The selection of tests for each study tasks will be determined either by the need to establish control data for a patient population currently being evaluated under a collaborative protocol, or to establish normative data on a test that will further expand our ability to investigate specific pathology/function for which no equivalent published normative data are available (e.g., otolith disease, auditory processing disorders). The specific tests that each participant will perform will be clearly indicated and described in the consent/assent documents and will be explained during the consent/assent process. Testing will be conducted during a single outpatient clinic visit with the exception of measures for which test-retest reliability is being investigated.

Outcome measures:

This is a normative data collection protocol designed to describe normal behavioral and physiologic auditory and vestibular function for the NIH research population. Outcome measures will vary from test to test and include one or more of the following: 1) response threshold, amplitude, latency, velocity, frequency response, and/or accuracy, 2) number and/or percent correct, 3) response repeatability, and 4) interaural response differences.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy adult volunteers:

* Healthy adults, aged 18-80 years
* Able to provide informed consent
* Normal hearing sensitivity, defined as pure-tone thresholds less than or equal to 25 dB HL, or when the pure-tone threshold exceeds 25 dB HL, it must be less than or equal to the median threshold for the appropriate gender- and age-based group, for 250-8000 Hz (Morrell et al, 1996, ISO-7029, 2000).
* No air-bone gaps in excess of 10 dB for 500-4000 Hz.
* Normal middle ear function as indicated by normal 226 Hz tympanograms bilaterally, defined as middle ear pressure between more or less 100 decaPascals, and peak compensated static compliance between 0.3-1.5 milliliters
* American English as a first language for those participating in study tasks evaluating auditory processing.
* Able to refrain from caffeine and alcohol for 48 hours before vestibular study sessions because both agents may modify the test results.

EXCLUSION CRITERIA:

* History of auditory and/or vestibular disorders (e.g., Meniere s syndrome, labyrinthitis).
* Evidence of active outer or middle ear disease or anomaly (e.g. otitis media, stenotic ear canal, otorrhea)
* History of chronic (fluid in middle ear for more than 4 months) or recurrent otitis media (more than 4 episodes of acute otitis media in one year)
* History of ear surgery other than PE tubes
* Current PE tubes
* History of treatment with ototoxic medications (e.g. cisplatin, aminoglycoside antibiotics)
* Unable to discontinue medications that can interfere with vestibular test results for the 48 hours immediately preceding a vestibular study session. These include any and all anti-dizziness medications (such as Antivert), prescription pain medications (such as Percocet), prescription headache medications (such as Imitrex), sleeping pills (such as Ambien), anti-seizure medications (such as Topamax), and/or antihistamines (such as Benadryl).
* Current diagnosis from the Diagnostic and Statistical Manual of Mental Disorders (DSM IV) of a psychiatric disorder or on medications for a psychiatric disorder in the past two years, including any or all antidepressants, anxiolytics, or psychostimulant drugs.
* Cognitive impairment as evidenced by a score <26 on the Montreal Cognitive Assessment (MoCA).
* Attention deficit hyperactivity disorder (ADHD) as evidenced by a score of greater than or equal than or equal to 4 on the Adult ADHD Self Report Scale (Kessler et al., 2005).
* History or diagnosis of a central nervous system disorder, including but not limited to:

  * Intracranial tumors
  * Cerebrovascular disease
  * Degenerative CNS disorder
  * CNS trauma
  * Encephalitis
  * Meningitis
* Current diagnosis of speech and/or language disorders, autism, auditory neuropathy, or auditory processing disorder; or in therapy for these disorders in past 2 years.
* Reduced visual acuity preventing ability to see the visual targets used for vestibular and balance testing as evidenced by corrected visual acuity worse than 20/25 on a Snellen chart for those participating in vestibular tasks.
* Ocular motor impairment preventing ability accurately follow the visual target used for calibration and/or ocular motor tasks for those participating in the vestibular tasks.
* Employees and staff of the Audiology Unit, Otolaryngology Branch, NIDCD.
* Reduced balance or postural instability as evidenced by a Timed Up and Go score greater than or equal to 11.1 seconds (Whitney et al., 2004) for adults <65 years of age and >12.6 seconds for adults 65-80 years of age (Shumway-Cook et al.,2000) and/or Activities-specific Balance Confidence Score <67% for those participating in vestibular study tasks.

Healthy children volunteers:

INCLUSION CRITERIA:

* Healthy children, aged 5 years-0 months to 17 years-11 months
* Normal hearing sensitivity, defined as pure-tone thresholds of 15 dB HL or better for 250-8000 Hz
* Normal middle ear function as indicated by normal 226 Hz tympanograms bilaterally, defined as middle ear pressure between more or less 100 decaPascals, and peak compensated static compliance between 0.2-1.5 milliliters
* American English as a first language for those participating in study tasks evaluating auditory processing.
* Ability to follow the verbal instructions and commands for study tests
* Able to refrain from alcohol and caffeine intake for 48 hours before vestibular study sessions because caffeine may modify the test results
* Weight greater than 40 pounds for those participating in vestibular tasks that include CDDP

EXCLUSION CRITERIA:

* History of auditory and/or vestibular disorders (e.g. Meniere syndrome, enlarged vestibular aqueduct).
* Evidence of active outer or middle ear disease or anomaly (e.g. otitis media, stenotic ear canal, otorrhea)
* History of chronic (fluid in middle ear for more than 4 months) or recurrent otitis media (more than 4 episodes of acute otitis media in one year)
* History of ear surgery other than PE tubes
* Current PE tubes
* History of treatment with ototoxic medications (e.g. cisplatin, aminoglycoside antibiotics)
* Unable to discontinue medications that can interfere with vestibular test results for the 48 hours immediately preceding a vestibular study session. These include any and all anti-dizziness medications (such as Antivert), prescription pain medications (such as Percocet), prescription headache medications (such as Imitrex), sleeping pills (such as Ambien), anti-seizure medications (such as Topamax), and/or antihistamines (such as Benadryl).
* Current diagnosis from the Diagnostic and Statistical Manual of Mental Disorders (DSM IV) of a psychiatric disorder or on medications for psychiatric disorder in the past two years, including any or all antidepressants, anxiolytics, or psychostimulant drugs.
* Cognitive impairment as evidenced by a standard score less than 85 on the Peabody Picture Vocabulary Test (Fourth Edition)
* Attention deficit hyperactivity disorder (ADHD) as evidenced by a score of greater than or equal to 6 on the SNAP IV
* History or previous diagnosis of a central nervous system disorder, including but not limited to:

  * Intracranial tumors
  * Cerebrovascular disease
  * Degenerative CNS disorder
  * CNS trauma
  * Encephalitis
  * Meningitis
* Current diagnosis of speech and/or language disorders or delays, autism, auditory neuropathy, or auditory processing disorder; or in therapy of these disorders in past 2 years.
* Reduced visual acuity preventing ability to see the visual targets used for vestibular and balance testing as evidenced by corrected visual acuity worse than 20/25 on a Snellen chart for those participating in vestibular study tasks.
* Ocular motor impairment preventing ability to see or accurately follow the visual target used for ocular motor tasks for those participating in the vestibular study tasks.
* Reduced balance or postural instability as evidenced by a Timed Up and Go score of greater than or equal to 9.4 seconds for those participating in vestibular study tasks.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers ranging in age from 5-80 years will be studied under this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-09-21 (Actual)

PRIMARY OUTCOMES:
Normative data for behavioral and physiologic auditory and vestibular function including 1) response threshold, amplitude, latency, velocity, repeatability, frequency response, accuracy, 2) percent correct and/or interaural response differences | Varies from test to test
  Outcome measures will vary from test to test and include one or more of the following: 1) response threshold, amplitude, latency, velocity, frequency response, and/or accuracy, 2) number and/or percent correct, 3) response repeatability, and 4) interaural response differences.

CONTACTS AND LOCATIONS:
Overall Officials: Gayla L Poling, Ph.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-DC-0152.html